CLINICAL TRIAL: NCT02718378
Title: A Phase I, Double-blind, Randomised, Placebo-controlled, Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Multiple Dosages of Estetrol in Healthy Men
Brief Title: Evaluation of Safety and Efficacy of Estetrol in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pantarhei Oncology B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PR3107
Record Dates: First submitted 2016-02-18; First posted 2016-03-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Prostatic Neoplasms
Keywords: safety; pharmacokinetics; pharmacodynamics; randomized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estetrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- No added active (Placebo Comparator): placebo without estetrol
  Interventions: Drug: placebo
- estetrol dose level 1 (Active Comparator): estetrol given in dose level 1
  Interventions: Drug: estetrol
- estetrol dose level 2 (Active Comparator): estetrol given in dose level 2
  Interventions: Drug: estetrol
- estetrol dose level 3 (Active Comparator): estetrol given in dose level 3
  Interventions: Drug: estetrol

INTERVENTIONS:
Drug: estetrol
  Arms: estetrol dose level 1; estetrol dose level 2; estetrol dose level 3
Drug: placebo
  Arms: No added active

SUMMARY:
The current study is designed as a phase Ib multiple dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of E4 in healthy men after daily oral administration for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male, age between 40 and 70 years (both inclusive);
* Good physical and mental health as judged by the Investigator determined by medical history, physical examination (including prostate palpation), clinical laboratory, vital signs and ECG recording;
* Body mass index between ≥ 18.5 and ≤ 30.0 kg/m2;
* Normal prostate-specific antigen (PSA) value (< 3.0 ng/mL);
* Non-vasectomized men must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication. Men who have been vasectomized less than 4 months prior to study start must follow the same restrictions as non-vasectomized men;
* Men must agree not to donate sperm from the first dose until 90 days after the last dose;
* Ability to communicate well with the Investigator and to comply with the requirements of the entire study;
* Willing to give informed consent in writing.

Exclusion Criteria:

* Any clinically significant abnormality following review of medical history, laboratory results, physical examination and ECG at screening as judged by the Investigator;
* Conditions or disorders that might affect the absorption, distribution, metabolism or excretion of any of the study drugs;
* Previous use of steroids within:

  * 8 weeks for oral preparations
  * 4 weeks for transdermal preparations
  * Any time for injections;
* Contraindications for steroids or estetrol;
* Prostate hyperplasia or micturition problems that suggest the presence of prostate hyperplasia;
* Presence of an active acute or chronic infection, including syphilis, HIV or viral hepatitis B and/or C (or previously treated);
* Treatment for any major psychiatric disorder in the previous 12 months or use of antidepressant medication before screening;
* Hypersensitivity to the active substances or to any of the excipients of the investigational product or placebo therapy;
* Use of probiotics (as present in dairy products, fortified foods etc.) during the 3 months before screening and during the clinical study;
* Use of one or more of the following medications:

  * Antihypertensive drugs
  * Present use or use within 30 days before the start of the study drug of the following drugs: aprepitant, bosentan, armodafinil, phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, glucocorticoids, topiramate, felbamate, rifampicin, clobazamechinacea; vemurafenib, non-nucleoside reverse transcriptase inhibitors, griseofulvin, ketoconazole, and herbal remedies containing Hypericum perforatum
  * Any medication (including over-the-counter products) within 14 days before first dosing except for occasional non-steroidal anti-inflammatory drugs (NSAIDs; e.g. ibuprofen); paracetamol is not permitted
  * Use of antibiotics;
* Administration of any other investigational drug within 3 months before first dosing;
* Loss of more than 400 mL blood during the 3 months before screening, e.g. as a blood donor, or intention to donate blood in the 3 months after completing the study;
* Subjects with a history of (within 12 months) alcohol or drug abuse or with a positive result at screening, for tests of:

  * alcohol intake
  * drug abuse;
* Currently smoking or smoked within the last 6 months before screening.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 28 days
  Changes from baseline measurements considered clinically significant by the Investigator will be reported as AEs.
Change from baseline in hormone levels | 28 days
  The serum concentrations of Follicle Stimulating Hormone (FSH), Luteinising Hormone (LH), Estradiol (E2), total testosterone and free testosterone levels (actual values as well as percentage change from pre-dose concentration) will be listed and summarized descriptively by treatment group.

SECONDARY OUTCOMES:
Change from baseline in haemostasis parameters | 28 days
  The relative change in Activated Protein C (APC)-resistance, prothrombin factor 1 + 2, D-dimer, free Tissue Factor Pathway Inhibitor (TFPI), antothrombin activity, protein S activity and angiotensinogen levels and the actual change from baseline will be calculated by treatment group.
Change from baseline in lipid parameters | 28 days
  The relative change in total cholesterol, triglycerides, High Density Lipoprotein (HDL) cholesterol, Low Density Lipoprotein (LDL) cholesterol, Lipoprotein A (Lp(A)) levels and the actual change from baseline will be calculated by treatment group.
Change from baseline in glucose levels | 28 days
  The relative change in glucose levels and the actual change from baseline will be calculated by treatment group.
Change from baseline in bone turnover markers | 28 days
  The relative change in osteocalcin, type I collagen telopeptide (CTX-1) and parathyroid hormone (PTH) and the actual change from baseline will be calculated by treatment group.
Change from baseline in sex-hormone binding globulin (SHBG) levels | 28 days
  The relative change in SHBG levels and the actual change from baseline will be calculated by treatment group.
Pharmacokinetic effect of estetrol | 28 days
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic effect of estetrol | 28 days
  Terminal elimination half-life (t1/2)
Pharmacokinetic effect of estetrol | 28 days
  Time to reach Cmax (tmax)
Pharmacokinetic effect of estetrol | 28 days
  Peak plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Tjeert Mensinga, MD, PhD, Principal Investigator — QPS Netherlands BV
Locations (1):
- QPS Netherlands BV, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Result] Phillips I, Shah SI, Duong T, Abel P, Langley RE. Androgen Deprivation Therapy and the Re-emergence of Parenteral Estrogen in Prostate Cancer. Oncol Hematol Rev. 2014 Spring;10(1):42-47. doi: 10.17925/ohr.2014.10.1.42. PMID 24932461
- [Result] Coelingh Bennink HJ, Holinka CF, Diczfalusy E. Estetrol review: profile and potential clinical applications. Climacteric. 2008;11 Suppl 1:47-58. doi: 10.1080/13697130802073425. PMID 18464023
- [Derived] Coelingh Bennink HJT, Zimmerman Y, Verhoeven C, Dutman AE, Mensinga T, Kluft C, Reisman Y, Debruyne FMJ. A Dose-Escalating Study With the Fetal Estrogen Estetrol in Healthy Men. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3239-3249. doi: 10.1210/jc.2018-00147. PMID 29931320